CLINICAL TRIAL: NCT00380484
Title: Short- and Long Term Growth in Children With Asthma Treated With Budesonide or Montelukast
Brief Title: Short- and Long Term Growth in Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children´s Clinic, Randers (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BKR-KNAST-06; EudractCT-nr 2006-003013-41
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; montelukast

ARMS (2):
- 1 (Experimental): Budesonide
  Interventions: Drug: Budesonide
- 2 (Active Comparator): Montelukast
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Budesonide — 200µg daily
  Arms: 1
Drug: Montelukast — 5 mg daily
  Other Names: Singulair
  Arms: 2

SUMMARY:
The purpose of this study is to assess if treatment with budesonide 200 microgram per day affects short- or long term growth in children with asthma

DETAILED DESCRIPTION:
When children with asthma are treated with inhaled corticosteroids there is a risk of systemic adverse events such as growth suppression. It has been reported that treatment with budesonide 200 microgram per day does not affect short term growth in children with asthma. The aim of the present study is to assess if an unaffected short term growth means that also long term growth will be unaffected.

Short and long term growth in asthmatic children treated with budesonide will be compared with the growth in asthmatic children treated with montelukast.

ELIGIBILITY:
Inclusion Criteria:

* age 6-11,
* prepubertal,
* asthma,
* normal weight and height,
* informed consent

Exclusion Criteria:

* treatment with systemic/inhaled/intranasal corticosteroids within the last week,
* major surgery within 4 weeks,
* usage of drugs that significantly inhibit CYP3A4

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Lower leg growth rate | one year
Height | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ole D Wolthers, Principal Investigator — Children's Clinic Randers
Locations (1):
- Children's Clinic Randers, Randers, Denmark